CLINICAL TRIAL: NCT01341691
Title: A 2 Week Single Blind Study to Evaluate Phosphate Binding of Chitosan Chewing Gum in Patients With Chronic Kidney Disease
Brief Title: Phosphate Binding of Chitosan Chewing Gum in Patients With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Denver Nephrologists, P.C. (Other)
Collaborators: CM&D Pharma, LTD (Unknown)
Responsible Party: Geoffrey A. Block, Denver Nephrologists, PC
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: CMD 006
Record Dates: First submitted 2011-04-23; First posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; K2CG chewing gum; phosphorus; saliva
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo 20mg (Placebo Comparator)
  Interventions: Other: chewing gum
- K2CG 60 mg extender (Active Comparator)
  Interventions: Other: chewing gum
- K2CG 60 mg (Active Comparator)
  Interventions: Other: chewing gum
- K2CG 20mg extender (Active Comparator)
  Interventions: Other: chewing gum
- K2CG 20mg (Active Comparator)
  Interventions: Other: chewing gum
- Placebo 60mg (Placebo Comparator)
  Interventions: Other: chewing gum

INTERVENTIONS:
Other: chewing gum — single piece of chewing gum containing specified amount of chitosan with or without extender chewed twice daily for 14 days

SUMMARY:
To determine the amount of phosphate recovered into 2 strengths of K2CG chewing gum in a modified formulation (with or without an extender) added to the gum core, in comparison to matching placebo gums.

DETAILED DESCRIPTION:
The current treatment for elevated serum phosphorus levels in chronic kidney disease (CKD) consists of dietary restriction of P and the provision of phosphate binders that act at the level of the intestinal absorption of phosphorus (P) when ingested with meals. This paradigm has proven to be inadequate to achieve normo-phosphatemia as indicated by elevated serum P levels in patients receiving renal replacement therapy.

Salivary phosphate levels are elevated in patients with CKD and salivary P represents a large source of otherwise hidden non-dietary phosphate that is easily absorbed and may contribute to persistent elevations in serum P despite standard therapy.

Savica et al performed a preliminary study, in a small population (n-13) of hyperphosphatemic patients receiving hemodialysis, phosphate restriction and phosphate binders, and given K2CG chewing gum 20 mg. The chewing gum was administered twice per day for 60 minutes during fasting periods (between meals) for 15 days. In addition to a significant reduction in salivary P, serum P was reduced by 2 mg/dL (31%) over the treatment period. Both salivary and serum P returned to baseline values after K2CG discontinuation. The authors concluded that adding salivary P binding to traditional phosphate binders could be a useful approach for improving treatment of hyperphosphatemia in patients receiving renal replacement therapy (RRT).

Given the public health importance of increased P levels in the general population and specifically in patients with chronic kidney disease, it is of great importance to evaluate the ability of a medical food such as K2CG to reduce elevated serum P levels. In patients with CKD receiving RRT it has been estimated that sustained control of serum P may result in an approximate 17% reduction in mortality.

The specific purpose of this study is to compare the total P recovered per piece of chewing gum with 20 mg and 60 mg versions of the reformulated K2CG with or without the extender in the gum core. Additionally, the unique P binding of the reformulated gum will be assessed in comparison with the total P entrapped per piece of chewing gum in the matching placebos.

Subjects will be assigned to one of 3 different groups as shown in the table below. The study will be a single blind study. Subjects will be blinded as to the strength/formulation of the chewing gum and the active/placebo assignment.

Group Active Chewing Week 1 Active Chewing Week 2 20 mg with extender 20 mg Placebo 20 Placebo 60 60 mg with extender 60 mg

Subjects will chew the K2CG gum of a single strength/formulation for 7 days (Active Chewing Week 1) twice a day (BID). K2CG gum must be chewed at least 60 minutes in fasting conditions. This will be followed by a second 7 days of chewing K2CG gum (Active Chewing Week 2) of a different strength/formulation as described above.

There will be no run-in period and no wash out period between Active Chewing Week 1 and Active Chewing Week 2.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years of age;
* The subject has voluntarily signed and dated the most recent informed consent form approved by an Institutional Review Board (IRB);
* The subject will, in the opinion of the investigator, be compliant with prescribed therapy;
* Subject must be able to communicate and be able to understand and comply with the requirements of the study;
* Subject must be prescribed a diet appropriate for patients with their stage of CKD and must be willing to avoid intentional changes in diet; and
* Subject must have completed the CMD002 clinical trial and is currently receiving hemodialysis.

Exclusion Criteria:

* Subject is receiving or has received an investigational product (or is currently using an investigational device) within 7 days prior to baseline;
* Subject has a known sensitivity to chitin or allergy to shellfish;
* Subject has a clinically significant infection requiring treatment with antibiotics (within 7 days prior to baseline);
* Subject has had an inpatient hospitalization within 7 days prior to baseline with the exception of hospitalizations related to vascular access procedures; In the opinion of the investigator, subject is unable to chew gum for 60 minutes; and
* Subject has an unstable medical condition which in the opinion of the investigator would compromise successful completion of the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Total phosphorus bound and entrapped per piece of chewing gum | 60 minutes
  Each subject will chew a single piece of chewing gum for 60 minutes, twice daily for 1 week and all gum is collected and analyzed individually.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrologists, PC
Locations (1):
- Denver Nephrologists, PC, Denver, Colorado, United States

REFERENCES:
- [Derived] Block GA, Persky MS, Shamblin BM, Baltazar MF, Singh B, Sharma A, Pergola P, Smits G, Comelli MC. Effect of salivary phosphate-binding chewing gum on serum phosphate in chronic kidney disease. Nephron Clin Pract. 2013;123(1-2):93-101. doi: 10.1159/000351850. Epub 2013 Jun 22. PMID 23797006